CLINICAL TRIAL: NCT05282615
Title: A Randomized, Controlled, Proof of Concept Trial of the Impact of Daily Use of The Emanate Tray Adjunct to Full Mouth Debridement Compared to Full Mouth Debridement Alone
Brief Title: Impact of Daily Use of The Emanate Tray Adjunct to Full Mouth Debridement Compared to Full Mouth Debridement Alone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emanate Biomedical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Emanate Tray 001
Record Dates: First submitted 2022-02-16; First posted 2022-03-16 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Wound Heal; Mouth; Wound; Periodontal Inflammation
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Treatment Group (Emanate Tray) (Experimental): Full mouth periodontal debridement + Emanate Tray (treatment group)
  Interventions: Device: Emanate Tray
- Control Group (No Intervention): Full mouth periodontal debridement alone (control group)

INTERVENTIONS:
Device: Emanate Tray — Emanate Tray, a personalized dental tray set (upper and lower) with PVA hydrogel containing 0.05% w/w chlorhexidine gluconate
  Arms: Treatment Group (Emanate Tray)

SUMMARY:
The study is a 56-day (8-week), randomized, controlled, examiner-blinded, parallel-design study of patients with existing Stage II or Stage III periodontitis. After eligibility determination, subjects will be randomized to the following groups:

* Group 1: Full mouth periodontal debridement + Emanate Tray (treatment group)
* Group 2: Full mouth periodontal debridement alone (control group)

Patients will be evaluated at Baseline and on Days 14, 28, and 56 for primary endpoint and at baseline and on day 56 post-treatment for secondary (efficacy) endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed, written informed consent prior to participation in any study-related procedures.
2. Good general health as evidenced by medical history.
3. At least 18 years of age at time of informed consent signature.
4. Minimum of 18 teeth, excluding third molars.
5. Generalized Stage II-III periodontitis with at least 8 teeth having interproximal clinical attachment level of ≥3 mm and a probing pocket depth of ≥4 mm and ≤7mm, distributed between mandible and maxilla, with at least 2 qualifying interproximal sites in each arch. Localized and not more than ≤6 sites with a PD of 8 mm is acceptable as long as the tooth with 8 mm pocket depth is not clinically diagnosed as hopeless tooth with suppuration or mobility Grade 3 or greater
6. Having ≥40 percent of sites with bleeding upon probing as a sign of inflammation
7. Willing to use prescribed oral hygiene procedures and products
8. Willingness to maintain their routine dental care
9. Willing to abstain from chewing gums, mouth rinses and whitening products for the study duration.
10. Ability and willingness to attend all study visits and comply with all study visits and all study procedures and requirements.
11. For women with reproductive potential, willingness to use highly effective contraception (e.g., licensed hormonal contraception, intrauterine device, or vasectomy in partner).

Exclusion Criteria:

1. Presence of orthodontic appliances (anterior fixed retainers are allowed as long as the qualifying teeth are not involved).
2. A soft or hard tissue tumor of the oral cavity.
3. Patients with heavy subgingival calculus.
4. Any dental condition that requires immediate treatment, such as carious lesions.
5. Dental implants will be excluded from study, but the patients will not be excluded if they are otherwise eligible
6. Periodontal treatment including SRP within the prior 6 months of enrollment.
7. Participation in any other clinical study within 30 days of screening or during the study.
8. Pregnancy or lactation.
9. Patients that are known to be hypersensitive to chlorhexidine gluconate, glycerin, polyvinyl alcohol, or ethylene vinyl acetate
10. Antibiotic therapy within the last month (30 days)
11. Current smoking (cigarette, cigar, e-cigarette, or marijuana) within 1 year of enrollment
12. Patients that have a history of testing positive for SARS-CoV-2 per patient's report (within last 10 days) or currently having lingering/long-term COVID symptoms.
13. Chronic use (≥3 times/week) of anti-inflammatory medications (e.g., non-steroidal anti inflammatory drugs, steroids). Low-dose aspirin, 81-162 mg is allowed.
14. Immunocompromised subjects (i.e., subjects with AIDS, pulmonary fibrosis, undergoing chemotherapy or radiation treatment etc.).
15. Diabetes Mellitus defined as a HbA1c > 6.5 per laboratory test results
16. Liver function test (aspartate aminotransferase [AST], alanine aminotransferase [ALT], alkaline phosphatase, and total bilirubin) levels equal to > 1.5 times the upper limit of normal
17. Serum creatinine levels equal to > 2 times the upper limit of normal
18. Any medical history or any concomitant medication that might affect the assessment of the study treatment or periodontal tissues, such as nifedipine, phenytoin (Dilantin), or anticoagulant medications (e.g., warfarin [Coumadin] etc.).
19. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 56 days
  The number and percentage of subjects who experience at least 1 treatment-emergent AE (TEAE) and the number and percentage of subjects who experience at least 1 TEAE within each specific system organ class (SOC) and preferred term (PT).

SECONDARY OUTCOMES:
To evaluate the primary efficacy-effect of Emanate Tray on bleeding and probing (BOP) | 56 days
  The % reduction in sites with BOP
To evaluate the effect of Emanate Tray on pocket depth (PD) reduction | 56 days
  The mean reduction in pocket depth at Day 56.
To evaluate the effect of Emanate Tray on clinical attachment level (CAL) | 56 days
  The mean reduction in clinical attachment level at Day 56.
To evaluate changes in plaque index (PI) | 56 days
  The mean reduction in amount of plaque at Day 56.

OTHER OUTCOMES:
To acquire preliminary information regarding the effect of Emanate Tray on inflammatory cytokine levels in gingival crevicular fluid (GCF) | 56 days
  The change in inflammatory mediator levels in GCF at Day 56 compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Forsyth Institute, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No